CLINICAL TRIAL: NCT01537263
Title: Ultrasound Perfusion Imaging After Aneurysmal Subarachnoid Hemorrhage
Acronym: PSAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Gunter Seidel, MD, MD, Professor of Neurology, Asklepios Kliniken Hamburg GmbH
Other Study IDs: 2371
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Aneurysmal Subarachnoid Hemorrhage; SAB; SAH; Ultrasound; Perfusion imaging
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound Perfusion Imaging: Patient with subarachnoid hemorrhage.
  Interventions: Device: Ultrasound Perfusion Imaging

INTERVENTIONS:
Device: Ultrasound Perfusion Imaging — Sonographic unit Phillips IU 22, 5ml SonoVue ultrasound contrast agent per examination, Duration: 1h

SUMMARY:
The purpose of this study is to examine wether delayed cerebral ischemia can be predicted by ultrasound brain perfusion imaging in patients with aneurysmal subarachnoid hemorrhage (SAH).

DETAILED DESCRIPTION:
The delayed cerebral ischemia is a main complication in patient with aneurysmal subarachnoid hemorrhage which causes neurological deficit. So far there is no reliable diagnostic tool to predict the appearance of cerebral ischemia.

The causal correlation between presence of cerebral vasospasm measured daily by transcranial Doppler sonography (TCD) and occurrence of cerebral ischemia detected by cranial computed tomography scan (CCT) is not finally verified.

First studies demonstrated that ultrasound perfusion imaging (UPI) allows the detection of perfusion deficits in middle cerebral artery infarction.

The purpose of our study is to evaluate the diagnostic and prognostic value of UPI to predict delayed cerebral ischemia. In our trial we compare parameters of UPI (b= rise rate, A= plateau of acoustic intensity) in patients with aneurysmal subarachnoid hemorrhage with results of follow-up cranial computed tomography scans (CCT), TCD results and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal subarachnoid hemorrhage, Hunt and Hess 0-5
* Informed consent
* Sufficient transtemporal acoustic window
* First examination within 48h after subarachnoid hemorrhage
* Minimum Age 18 years

Exclusion Criteria:

* Contraindication against computed tomographic scan
* Incompatibility against SonoVue™
* Acute respiratory distress syndrome
* Uncontrollable hypertensive crisis
* Severe pulmonary disease(pulmonary hypertension > 90 mmHg)
* acute severe cardiac insufficiency (New York Heart Association IV)
* known right-left-shunt
* pregnancy and breastfeeding
* Substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change of perfusion | Baseline, Day 5
  Detection of hypoperfusion (defined by 50% or more reduction in beta-value of comparing day 1. with day 5.) in one or more of four regions in one or both hemispheres before the detection of delayed ischemia after SAH in CCT.

SECONDARY OUTCOMES:
Correlation between perfusion parameters, clinical course and flow velocities | Day 1 to 90
  Correlation between perfusion parameters (beta- and A-value), clinical course (National Institute of Health Stroke Scale - NIHSS) and flow velocities in the middle and posterior cerebral artery from day 1 to day 90.
Change of Perfusion | Baseline, Day 5
  Detection of hypoperfusion (defined by 50% or more reduction in A-value of comparing day 1. with day 5.) in one or more of four regions in one or both hemispheres before the detection of delayed ischemia after SAH in CCT.

CONTACTS AND LOCATIONS:
Overall Officials: Günter Seidel, MD, Professor of Neurology, Study Director — Asklepios Kliniken Hamburg GmbH
Locations (1):
- Department of Neurology, Asklepios Hospital North, Hamburg, Hamburg, Germany